

# **EIRB Protocol Template (Version 1.1)**

# 1.0 General Information

| "Please enter the full tit | ie of your study. | |
|---|---|---|
| Does self-efficacy predict i<br>during initial entry training? | injury and training outcomes among U.S. Military Academy cadets ? | |
| *Please enter the Protoc | col Number you would like to use to reference the protocol: | |
| 22KACH007 * This field allows you to enthis protocol. | nter an abbreviated version of the Protocol Title to quickly identify | |
| Is this a multi-site study | (i.e. Each site has their own Principal Investigator)? | |
| No | | |
| Does this protocol involv | ve the use of animals? | |
| Yes • No | | |
| 2.0 Add Site(s) | | i I |
| 2.1 List sites associated v | with this study: | |
| Department Department Department Department A | rmy Community Hospital (KACH) | |
| 3.0 Assign project | personnel access to the project | |
| 3.1 *Please add a Princip | eal Investigator for the study: | |
| Kreisel, Brian Robert, Doctora | ate of Science MAJ | |
| Select if applicable D Student | D Site Chair | |
| Resident | Fellow | |
| 3.2 If applicable, please s | select the Research Staff personnel: | |
| A) Additional Investigators | | |
| Benedict, Timothy <b>M</b> , PhD, D | PT LTC | |
| Associate Investigator Casper, Preston C, Doctorate | | |
| Gasper, Freston G, Doctorati | о пі і пузісаі і петару 🗀 | |

| Associate Investigator | | 1 | Ī |
|---|---|---|---|
| Crowell, Michael SCOTT, DPT, DSc LTC | | | |
| Associate Investigator | | | |
| Dummar, Max Ken | | | |
| Associate Investigator | | | |
| Francis, Matthew W, DPT MAJ | | | |
| Associate Investigator | | | |
| Kuwik, Paul ANDREW, DPT | | | |
| Associate Investigator | | | |
| Scott, Kelly Maureen | | | |
| Associate Investigator | | | |
| Associate investigator | | | |
| B) Research Support Staff | | | |
| Miller, Erin Marie, PhD | | | |
| Research Coordinator | | | |
| 3.3 *Please add a Protocol Contact: | | , , | |
| Benedict, Timothy M, PhD, DPT LTC | | | |
| Kreisel, Brian Robert, Doctorate of Science MAJ | | | |
| Scott, Kelly Maureen | | | |
| The Protocol Contact(s) will receive all important system no Investigator. (i.e. The protocol contact(s) are typically either Principal Investigator themselves). | | | |
| 3.4 If applicable, please select the Designated Site A | Approval(s): | <del></del> | |
| Haley, Chad Allen | | | |
| Department Chair | | | |
| 7 | | | |
| Add the name of the individual authorized to approve and (e.g. the Site Chair). | sign off on this protocol from your Site | | |
| 4.0 Project Information | | | |
| | | | 1 |
| 4.1 * What department(s) will be associated with the | his protocol? | | |
| II . | | | |
| Physi_l <u>Thernpy</u> l | | | |
| 4.2 * Has another IRB/HRPP reviewed this study or | _ | is study? | If |
| Yes, answer the questions according to the IRB | | | |
| Yes, answer the questions according to the IRB | | | |
| O Yes G No | | | |
| | Determination | | |
| O Yes G No | Determination | | |
| O Yes G No IRB Name Review Date | Determination | | |

| @ Yes O No | |
|---|---|
| 4.4 What type of research is this? | |
| I?Biomedical Research Clinical trial (FDA regulated) Behavioral Research Clinical trial (FDA regulated) | |
| 4.5 Are you conducting this project in pursuit of a personal degree? | |
| @Yes O No | |
| * Is this human subjects research? (As defined by 32 CFR219) Human subject means individual about whom an investigator (whether professional or student) conducting re (i) Obtains information or biospecimens through intervention or interaction with the is uses, studies, or analyzes the information or biospecimens; or (ii) Obtains, uses, studies, analyzes or generates identifiable private information or ide biospecimens. | esearch:<br>ndividual, and |
| ® Yes O No | |
| 4.8 * Do you believe this human subjects research is exempt from IRB review? | |
| O Yes @ No | |
| 5.0 Personnel Details | |
| 5.1 List any Research Team members without EIRB access that are not previously protocol: | entered in the |
| Norecords have been added | |
| 5.2 Will you have a Research Monitor for this study? | |
| O Yes<br>@ No<br>O N/A | |
| 6.0 Data/Specimens | |
| 6.1 Does the study involve the use of existing data or specimens only (no interaction with human subjects)? | on |

# 7.0 Funding and Disclosures

| 7.1 | Source | of Funding: | | | | | | |
|---|---|---|---|---|---|---|---|---|
| п | Funding So | urce | Funding Type | | Amount | | | |
| ſ | No records | have been added | 1 | | | | | |
| T | otal amoun | t of funding: | | | | | | |
| 7.2 | _ | - | vestigator(s) hav<br>or(s), product(s) | | | | | |
| 0 | Yes $0$ | No | | | | | | |
| If | Yes, comp | lete and attach C | Conflict of Interest | forms for all key | personnel | | | |
| 8.0 | | y Locations | | | | | | |
| 8.1 | Is this a | a collaborative | or multi-site stu | dy? (e.g., are t | here any ot | her institutio | ons involve | d?) |
| 0 | Yes @ | No | | | | | | |
| 8.2 | Study F | acilities and Lo | cations: | | | | | |
| | Institution | Site Name | Site Role | FWA or DoD<br>Assurance<br>Number | Assurance<br>Expiration<br>Date | Is there an agreement? | IRB Reviewi<br>for Site | ng |
| | Army | Keller<br>Army<br>Community<br>Hospital | Performance<br>site | 000029527 | 10/28<br>/2025 | | NM0<br>IRB | |
| O | ther: | | | | | | | |
| | Other<br>Institution | | FWA or DoD<br>Assurance<br>Number | FWA or Do<br>Expiration<br>Date | Is the | | B Reviewing<br>r Site | |
| _ | | have been added | | | | | | |
| 8.3 | Are the | re international | sites? | | | | | |
| | | ational approval<br>ntext has been co | documents, if app | licable, when pr | ompted. Not | te: Ensure loc | al | |
| 0 | Yes <i>Gi</i> | No | | | | | | |

| 8.4 Is this an ocoNus (Outside Continental United States) study? |
|---|
| <b>0</b> Yes @ No |
| Select the area of responsibility: |
| Have you obtained permission from that area of responsibility? (This is a requirement prior to study approval) |
| O Yes O No |

9.0

# Study Details

| 9.1 Key Words: |
|---|
| Provide up to 5 key words that identify the broad topic(s) of your study self-efficacy; musculoskeletal injury; tactical performance; initial-entry training |
| 9.2 Background and Significance: |

Include a literature review that describes in detail the rationale for conducting the study. Include descriptions of any preliminary studies and findings that led to the development of the protocol. The background section should clearly support the choice of study variables and explain the basis for the research questions and/or study hypotheses. This section establishes the relevance of the study and explains the applicability of its findings

Since World War I, U.S. Army leaders have faced a challenging conundrum: conduct training tough enough to prepare Soldier for warfare's physical and mental demands without causing so many injuries that units become non-deployable (East, 2013). The steady decline in physical activity levels and increases in overweight and obese adolescents (Center for Disease Control and Prevention /Division of Adolescent, 2020) has continued to widen the physical readiness gap between the general population and military physical demands (Alemany et al., 2021). This disparity increases the difficulty to train physically capable recruits without injuring those who are less fit.

Despite efforts to improve Soldier readiness, as many as 58,400 Soldiers were not capable to deploy in April 2020, which is equivalent to 13 Brigade Combat Teams (Department of the Army, 2020). More than half (31,500) were due to either temporary or long-term physical limitations, including musculoskeletal injuries (MSKIs). MSKIs are the leading cause of nondeployability, lost duty days (LDD), medical encounters, military discharge, and disability (Molloy, Pendergrass, Lee, Chervak, et al., 2020; Roy et al., 2021). In 2018 the U.S. Army spent \$434 million in direct medical costs alone to treat MSKIs (Molloy, Pendergrass, Lee, Chervak, et al., 2020).

Ironically, the leading causes of MSKIs are same activities that leaders deliberately conduct to develop physical resilience: running, foot marching, other physical fitness training activities (besides running) and work-related tasks (Roy et al., 2021). Although physical training results in the highest number of total injuries, obstacle courses and ruck marching have greater injuries per exposure (Lovalekar et al., 2021). Other common causes of MSKIs include overexertion, falls/slips, and accidental injury (Army Public Health Center, 2021).

Lower back injuries are a common occurrence in athletes and sports programs. They are especially common in sports in which athletes train strength and power movements, such as powerlifting and weight lifting (Bengtsson, 2018; Reichel, 2019; Stromback, 2018). Tactical athletes-referring to firefighters, police officers, and military servicemembers- report similar prevalence of low back pain (LBP), often due to heavy equipment worn or carried for their jobs (Roy, 2021). In the US military, musculoskeletal (MSK) injuries are highly prevalent and costly in lost duty days, depleted readiness to deploy, and medical expenses (Grimm, 2019; Teyhen, 2018).

Researchers have identified multiple physical and behavioral MSKI risk factors including prior injury, female gender (Hearn et al., 2021; Kucera et al., 2016), high or low BMI (Lovalekar et al., 2021; Rappole et al., 2017), history of smoking, low aerobic endurance (Molloy, 2016; Rappole et al., 2017),

and (to a lesser extent) muscular strength and endurance (Jones et al., 2017). Unit leaders and military trainers have used these study outcomes to develop injury prevention and training program including physical fitness programs, MSKI risk screening and leader education with mixed results (Canham-Chervak et al., 2015; Lovalekar et al., 2021; Molloy, Pendergrass, Lee, Hauret, el al., 2020; Terry et al., 2018).

These epidemiological and correlational studies summarize the dilemma: Soldiers with prior injury and lower fitness levels tend to get injured (again) while training to improve their physical fitness. It is possible that other modifiable risk factors exist that, if trained, do not carry such high injury risk.

The Army's new mandatory fitness test-Army Combat Fitness Test (ACFT)- is a comprehensive assessment of strength, power, speed, and endurance, and represents a dramatic shift from the previous fitness lest that primarily evaluated soldiers' endurance. One event of the ACFT is a three-repetition maximum deadlifl. The addition of a required deadlifl strength test has raised concern amongst servicemembersand healthcare workers about the risk of injury (Hauschild, 2019; Kind, 2019). The Army doctrine specifies the purpose of testing this event is to evaluate a soldier's lower body and core strength to safely lift heavy equipment, and the graders are instructed to not permit any lumbar flexion during the deadlift. (Army Field Manual 7-22).

Many coaches and physical therapists agree that lumbar flexion should not be permitted during a deadlifl (Nolan, 2019; Sjoberg, 2020; Spencer, 2015) however the majority of the research supporting this is based on empirical data derived from biomechanical or cadaver studies (Arjmand, 2005; Cholewicki, 1991; Dolan, 1994; Faber, 2009; Gallagher, 2012; Potvin, 1991; von Arx, 2021; Wade, 2014). There is some debate amongst researchers regarding the importance of avoiding lumbar flexion for injury back injuries during a deadlift (Adams, 1986, 1994; Beach, 2018; Spencer, 2015).

Alberto Bandura (1977) introduced self-efficacy as one's confidence to perform a specific task. In behavioral psychology, this concept helps patients and clinicians establish a therapeutic path by accomplishing individualized, increasingly difficult tasks (Bandura, 1977). Multiple subsequent publications have proposed positive relationships between self-efficacy and self-regulation (Bandura, 1982), performance (Bandura, 1982; Feltz et al., 2008), goal-setting (Brinkman et al., 2020) and motor learning (Beattie et al., 2014).

Performance effects resulting from the messages provided to athletes shouldn't be ignored, and this is referred to as placebo (has a perceived positive effect) or nocebo (has a perceived negative effect (Horvath, 2021). Theconcept of performance decline after negatively-perceived stimulus has a less robust presence in the literature than placebo effects, though this is evolving. Numerous recent studies have now documented the significant detriments to physical performance when subjects are exposed to negative or potentially threatening information (Cook, 2012; Corsi, 2019; Emadi Andani, 2015; Horcajo, 2019; Jackson, 2005; Pollo, 2012; Zech, 2019).

To our knowledge, there are no longitudinal studies evaluating the risk of injury from deadlifting with a flexed lumbar spine resulting in no clear evidence that a flexed spine is a risk factor for injury. However, it is well documented that information related to potential threat (nocebo) can adversely affect physical performance. Our research aim is to determine if cautionary information about the risk of spine injury harms performance on a maximum strength test compared to a message of spine resiliency. The cautionary education is similar to standard information provided to many servicemembers before the start of an ACFT or a maximum deadlift.

#### 9.3

#### Objectives/Specific Aims/Research Questions:

Describe the purpose and objective(s) of the study, specific aims, and/or research questions /hypotheses

- 1. Determine if general self-efficacy is a predictor of injury during Cadet Basic Training(CBT) by performing a Kaplan-Meier Survival Curve of a single self-efficacy assessment (Cadet General Self-Efficacy Assessment) and injury occurrence using the Defense Medical Surveillance System (DMSS), Cadet Illness and Injury Tracking System (CIITS), Armed Forces Health Longitudinal Technology Application (AHLTA) and a follow-up self-reported injury assessment.
  - 1. Independent Variable: Cadet General Self-Efficacy score

- 2. Dependent Variables: Injury report according to CIITS, AHLTA, DMSS, sick call report or self-reported
- 2. Determine if task-specific self-efficacy is a predictor of injury during specific CBT events by performing a Kaplan-Meier Survival Curve, a single assessment of cadet task-specific self-efficacy and injury occurrence using DMSS, CIITS, AHLTA and a follow-up self-reported injury assessment.
  - 1. Independent Variable: Cadet Task-Specific Self-Efficacy score
  - 2. Dependent Variables: Injury report according to DMSS or self-reported
- 3. Determine if general self-efficacy is a predictor of performance during CBT by performing a multivariate regression between a single self-efficacy assessment and multiple measures of performance during CBT including 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) raw or calculated score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events.
  - 1. Independent Variable: Cadet General Self-Efficacy score
- 2. Dependent Variables: performance outcome by event- 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events.
- 4. Determine if task-specific self-efficacy is a predictor of performance during CBT by performing a multivariate regression between a single (or multiple) assessments of cadet task-specific self-efficacy, and multiple measures of performance during CBT including 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) raw or calculated score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events.
  - 1. Independent Variable: task-specific self-efficacy scores
- 2. Dependent Variables: performance outcome by event including 1) successful completion (pass /fail), 2) basic rifle marksmanship qualification score, 3) 12-mile road march outcome (pass/fail), 4) Army Combat Fitness Test (ACFT) score, 5) land navigation score, 6) swimming assessment outcome (pass/fail) and 7) any other individually-graded events.
- 5. After completing CBT, determine which sources of self-efficacy ((1) enacting mastery experiences, 2) vicarious experiences, 3) verbal persuasion, 4) physiological state, 5) affective state, 6) mental imagery) were the most influential on cadets' self-efficacy throughout CBT specific tasks by conducting a Chi-square test.
  - 1. Independent Variable: reported level of influence of each (6) source of self-efficacy.
- 2. Dependent Variables: performance outcome by event including 1) successful completion (pass /fail), 2) basic rifle marksmanship qualification score, 3) 12-mile road march outcome (pass/fail), 4) Army Combat Fitness Test (ACFT) score, 5) land navigation score, 6) swimming assessment outcome (pass/fail) and 7) any other individually-graded events.
- 6. Determine the effect of low back pain education (cautionary vs resiliency) on deadlift performance (weight lifted).

We will analyze this with MDL weight lifted as the dependent variable (one-way ANOVA), with a planned comparison analysis if significant differences are found between groups.

7. Determine the degree of confidence cadets have in their ability to succeed at the MDL both before and after the education and MDL

We will analyze if there is a main effect of time in the pre-to-post self-efficacy scores with a paired ttest. We will use multiple regressions to analyze the impact of self-efficacy scores on MDL performance.

- 8. Determine the effect of low back pain education (cautionary vs resiliency) on deadlift self-efficacy. We will analyze change scores with one-way ANOVA with planned comparisons between groups if ANOVA is significant.
- 9. Determine the effect of low back pain education (cautionary vs resiliency) on perceived spine vulnerability on a deadlift.

We will analyze change scores with one-way ANOVA with planned comparisons between groups if ANOVA is significant.

| 9.4 | Study Design: |
|-----|---------------|

Describe study design in one to two sentences (e.g., prospective, use of existing records/data /specimens, observational, cross-sectional, interventional, randomized, placebo-controlled, cohort, etc.). Specify the phase - Phase I, II, III, orIV- forFDA-regulated investigational drug research

Tl1is study willbe a randomized controlled trial with parallel design and I:I allocation ratio. We planto use cluster randomization. We willhave three groups- control, cautionary, resiliency (Jackson, 2005).

9.5 Target Population:

Describe the population to whom the study findings will be generalized

U.S. Military Academy Cadets

#### 9.6 Benefit to the DoD:

State how this study will impact or be of benefit to the Department of Defense

Researchers inside and outside of the military have also found that self-efficacy predicts both performance and is negatively correlated with MSKI (Gruber et al., 2009; Samuels et al., 2010). In a study on Navy SEAL training resilience, researchers found that successful graduation was related to physiological markers of resilience (Ledford et al., 2020). However, few studies have investigated the combined effects of physical, behavioral and psychological factors on predicting MSKIs.

Cadet basic training (CBT) at the United State Military Academy (USMA) is a 7-week initial-entry training event that physically and psychologically prepares cadets to become officers. It includes similar training events and physical demands as other initial-entry military courses such as a 12-mile foot march with 35 lbs., physical training including running multiple days per week, weapons familiarization, and basic tactical training. The injury risk factors for cadets attending CBT are similar to trainees attending U.S. Army Basic Combat Training and regular military training even though injury incidence is lower (Hearn et al., 2021). Identifying self-efficacy as an injury risk factor is the first step to designing and implementing injury prevention measures. The purpose of this study is to investigate relationships between performance, MSKI and self-efficacy alone and in combination with other MSKI risk factors in USMA cadets participating in CBT.

There is currently an emphasis in Army Doctrine (FM 7-22) on form/technique for events on the ACFT, especially the maximum deadlift (MDL) and the prevention of lower back injuries. The rationale behind this is due to the perception that breakdowns in form during the deadlift lead to injuries, however, the research does not support this. Specifically, the research is unclear regarding the position of the spine while deadlifting- neutral vs flexed. Our results could impact future DoD publications regarding technique on the MDL and de-emphasize the role of a rounded spine as a safety concern.

The researchers hypothesize that self-efficacy (general and task-specific) will be positively correlated with successful completion and performance and negatively correlated with MSKI risk during CBT. The researchers will also explore the relationship between self-efficacy and other known injury risk factors. Furthermore, we hypothesize that such beliefs about the vulnerability of the spine to injury might contribute to future disabling beliefs about back pain. This research marks an important step in investigating the role of beliefs about the back and readiness.

10.0

# Study Procedures, Data Management, and Privacy

#### 10.1 Study Procedures:

Describe step-by-step how the study will be conducted from beginning to end

Phase I: Consent and Self-Efficacy Assessment

All new cadets are eligible to participate in this study and willreceive verbal and written study desc1iption dming the first or second week of cadet basic training. Immediately after consenting to pat1icipate, they will complete the study demographic data information ai1d the Cadet Basic Training Projective Performance

Invent01y, which assesses self-efficacy measured prospectively via questionnaire on a IO-point Likert scale from 1 (no confidence) to 10 (folly confident) for overall perfonnance dming cadet basic training, marksmanship/live fire training, mck marching 12 miles, land navigation, swimming, and the Anny Combat Fitness Test. It will also assess for any recent injuries and whether the injmy is cuffently hinde1ing them.

#### Phase 2: Injury Smveillance During Cadet Basic Training

TI1e researchers will monitor the Cadet Injury and Illness Tracking System (CIITS), Aimed Forces Health Longitudinal Technology Application (AHLTA) and the Defense Medical Strueillance System (DMSS) up to weekly to track injmies for the duration and for up to 9 weeks afte1wards. They will classify injuries as by diagnosis, region, and impact on training ("not injured" (1), "injured-not limited" (2), "injured-modified training" (3) and "injured-limited" (4)). Cadets will initially be defaulted as "not injured" (1). They will also complete the Single Assessment NIIIlleric Evaluation (SANE), rating their cuffent ability level on a scale of 0-100% with regards to their injury.

#### Phase 3: Maximum Deadlift and Low Back Pain Education

TI1e randomized control element of this study will occur before and during the maximum deadlift (MDL) of the Aimy Combat Fitness Test. At the start of cadet basic training, researchers will randomly allocate each company of cadets into a group receiving a cautionary message regarding risk of spine injmy, a group receiving a reassming me.ssage of spine resiliency, and a group receiving no education prior to the MDL. This education will include infonnation about the lumbar spine as it relates to a deadlift. The researchers will administer this education shortly prior to cadets taking the MDL. Cadets, test graders, and data analysts will all be blinded to group allocation. The researchers will collect MDL scores from each group and explore relationships between group assignment and MDL performance.

Because the study is deceptive, all subjects will be provided a handout with best-evidence summary statements on how to maintain a healthy back as a cadet and beyond. All patiicipants will be given this infonnation, debriefed and provided an opportunity to speak with a licensed physical therapist about any concerns they might have about their back or lifting for the deadlift at a later date.

#### Phase 4: Perfo1mance Outcomes

TI1e researchers will receive cadet perfonnance outcomes from the Department of Militaiy Instruction (DMI) and the Department of Physical Education (DPE). At a minimum, this will include overall outcome (pass/fail) and Aimy Combat Fitness Test (ACFT) raw ai1d calculated scores. If available, this will also include marksmanship score, live fire score, land navigation score, swim test pass/fail outcome, road maid1pass/fail outcome. TI1e reseai-chers will enter this data into the reseai-ch database.

Phase 5: Post-Cadet Basic Training Injmy Questionnaire and Self-Efficacy Sources

After cadet basic training, the cadets will complete an electronical injmy assessment questionnaire.

This v.ri.11 ensm·e that any cadets who coped with an injmy or self-modified training (such as pe1fonning at a lower level) ai·e also captured. This questionnaire will also classify the injuries according to the saine classification system as in phase 2. Thecadets will also answer questions related to the sources of confidence dming task-specific CBT events.

#### 10.2 Data Collection:

Describe all the data variables, information to be collected, the source of the data, and how the data will be operationally measured.

Cadet Demographics: Age, gender, height, weight, USMA Preparatory School attendance, intended athletics participation, intended USMA performance

Injury Questionnaire: Recent injury information (within last year), still effecting performance, and Single Assessment Numeric Evaluation (SANE), and after-cadet basic training injury presence, region, and limiting classification

Self-Efficacy: Overall Cadet Basic Training performance, marksmanship, buddy team live fire, swimming 150 yards, ruck marching (load carriage), ACFT, deadlift, land navigation

Maximum Deadlift (MDL) performance: Measured by the amount of weight successfully lifted during the ACFT.

Reported Self-Efficacy Source: Measured on the post-CBT survey using Qualtrics. The cadets will rank-order commonly cites sources of self-efficacy from most to least influential. The options will include commonly-cited self-efficacy sources: physiological state, previous experiences, affective state, mental imagery, vicarious experiences, and verbal persuasion.

| verbal, hard copy and electronic? | |
|---|---|
| ® Yes O No | |
| 10.4 Review the definitions below and respond to the following two questions. If you are answers, email DHA.PrivacyBoard@mail.mil for assistance. The Military Health Syst defined as all DoD health plans and DoD health care providers that are organized un management authority of, or in the case of covered individual providers, assigned to the Defense Health Agency (DHA), the Army, the Navy, or the Air Force MHS wor are employees, volunteers, trainees, and other persons whose conduct, in the perfet for the MHS, is under the direct control of the MHS, whether or not they are paid by business associates are persons or entities that provide a service to the MHS and rehealth information (PHI) to provide the service. | tem (MHS) is nder the or employed by, which was been decided by the contract of work the MHS. MHS |
| Are you an MHS workforce member? | |
| @ Yes, I am an MHS workforce member | |
| No, I am not an MHS workforce member | |
| Are you an MHS business associate? | |
| Yes, I am an MHS business associate | |
| @ No, I am not an MHS business associate | |
| 10.5 Have you consulted with an MHS data expert to determine the data elements requir | ed for your study? |
| Consulting with a data expert often saves time later in the compliance process because the data expert can advise on the data available in the numerous MHS information systems, the quality of that data and the methods for encrypting and collapsing data. To schedule a consult with an MHS data expert, send an email to: (DHA.PrivacyBoard@mail.mil) | |
| Yes, then complete the questions below according to the data consult | |
| ${f @}$ No, then complete the questions below according to the best of your knowledge | |
| 10.6 Indicate how you will request data from the MHS. Select all that apply. | |
| Talking with MHS health care providers or MHS health plans about specific research participants | |
| D Obtaining MHS hard copy records specific to research participants | |
| Obtaining data from an MHS information system(s) | |
| 10.7 If youare obtaining data from an MHSinformation system(s), indicate whether you data extract or whether you plan to access an MHS information system directly to | |
| A data extract is when the MHS or a contractor provides the data set directly to the researcher. When receiving a data set through data extract, the researcher may indicate whether the data elements should be provided as is, encrypted or collapsed. In contrast to a data extract, access to an information system means that the researcher may directly access an MHS information system and create a data set for the research study | |
| Data Extract | |
| P' Access | |
| 10.8 Doyouintend to request de-identified data from the MHS in your research study? | 1 |
| There are different two methods for de-identifying data pursuant to HIPAA: 1) Safe Harbor Method: Removing all of the identifiers listed in Table 1 below, provided that the researcher does not have actual knowledge that the remaining data can be used alone or in combination with other information to identify the individual who is the subject of the information. | |

| · | ppropriate knowledge of and experience with generally iples and methods for rendering information not the data is not individually identifiable | |
|---|---|---|
| O Yes ® No | | |
| 10.9 Indicate the MHSinformation | system(s) from which you will seek to obtain data | |
| | tains the data elements you need, refer to the Guide for or request guidance from an MHS data expert at: <b>DHA.</b> | |
| • | s systems. If the system from which you seek to obtain of the system in the "Other MHS Systems" category below | |
| HS Information System | Requesting Data | |
| I AHLTAI | <u>I</u> = IYesl | |
| <u>DMss</u> I | <u>I</u> = IYesI | |
| TMoosl | <u>I</u> = <u>IYes</u> l | |
| Pll -Only Systems: | • | |
| M HS Information System | questing Data | |
| No records have been added | | |
| De-Identified Data & Other System | e. | |
| | 3. | |
| In formation System | Requesting Data | |
| In formation System Other MHS System (May include PII PHI) | Requesting Data | |
| Other MHS System (May include PII | Requesting Data | |
| Other MHS System (May include PII PHI) | and/or I <u>Yes</u> | |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy | and/or I <u>Yes</u> | |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or o | and/or I <u>Yes</u> | es |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or o outside of the MHS, includir | and/or IYes | es |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or o outside of the MHS, including | and/or IYes | es |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or o outside of the MHS, including O Yes, will merge data ®No, will not merge data 10.11 Indicate the data elements also | and/or IYes | d |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or or outside of the MHS, including the MHS, including the MHS, will merge data ®No, will merge data 10.11 Indicate the data elements all members of the research partinformation systems. If you will merge data, also it relatives, employers, or hour | and/or IYes | d<br>HS |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or or outside of the MHS, including the MHS, including the MHS, will merge data ®No, will merge data 10.11 Indicate the data elements all members of the research parainformation systems. If you will merge data, also is | and/or IYes IYes Iyes Iyes | d<br>HS |
| Other MHS System (May include PII PHI) List other system here: Cadet Illness and Injury Tracking Sy (CITTS) 10.10 Do you intend to merge or or outside of the MHS, including the MHS, including the MHS, will merge data ®No, will merge data 10.11 Indicate the data elements all members of the research partinformation systems. If you will merge data, also it relatives, employers, or hour | and/or IYes IYes Iyes Iyes | d<br>HS |

| 2. Postal address<br>with only town,<br>city, state and zip<br>code | | | С |
|---|---|---|---|
| 3. Postal address with all geographic subdivisions smaller than a state, including street address, city, county, precinct, zip code and their equivalent geocodes, except for the initial three digits of a zip code if, according to the current publicly available data from the Bureau of Census: 1) the geographic unit formed by combining all zip codes with the same three initial digits contains more than 20,000 people; and 2) the initial three digits of a zip code for all such geographic units containing 20,000 or fewer people is changed to 000 | | | 0 |
| 4. Dates including all elements (except year) directly related to an individual, including birth date, admission date, discharge date, and date of death | n | [J | - |
| 5. Ages over 89 and all elements of dates (including year) indicative of such age, unless you will only request a single category of "age 90 or older" | 0 | 0 | Ci |
| 6. Telephone numbers | | [1] | r |

| | n | n | r |
|---|---|---|---|
| 8. Electronic mail addresses | n | rJ | r |
| 9. Social Security<br>numbers (SSNs) | | n | r |
| 10. Medical record numbers | | 0 | r |
| 11. Health plan beneficiary numbers | n | rJ | n |
| 12. Account numbers | D | D | С |
| 13. Certificate<br>/license numbers | D | D | С |
| 14. Vehicle identifiers and serial numbers, including license plate numbers | r1 | r:"J | r |
| 15. Device identifiers and serial numbers | | D | С |
| 16. Web Universal<br>Resource Locators<br>(URLs) | | | D |
| 17. Internet Protocol (IP) address numbers | D | D | С |
| identifiers, including finger and voice prints | | D | С |
| 19. Full-face photographic images and any comparable images | n | D | r |
| 20. Any other unique identifying number, characteristic, or code (Diagnosis, | n | 0 | r |

| DEERS ID, EDIPI,<br>Rank) | |
|---|---|
| If you are obtaining SSNs, provide a justification as to why and explain why a substitute cannot be used | |
| 10.12 Doyoubelieve it is possible for the MHS data to become identifiable because of trian small cell size, or any unique data element(s)? | gulation, a |
| Triangulation means using different data elements that are not themselves identifiable but that when combined can be used to identify an individual. For example, triangulation would use rank and race together to determine the identity of an individual with a particular health condition. | |
| Small cell size means that there is only a small number of eligible individuals that satisfy the category description. Guidance for acceptable cell size is available from the Centers for Medicare and Medicaid Services. For example, the rank category of four star generals with a particular diagnosis may be less than 30, so the rank category may need to be expanded to include lower ranks. | |
| A unique data element includes any unique features that are not explicitly enumerated in the categories of data in rows 1 - 20 of the table above (in Section 10.10), but that could be used to identify an individual. Unique data elements include characteristics that are not themselves identifying, such as the rank of general or admiral, or a race or gender, but within the context of other information could be identifiable. | |
| <b>0</b> Yes, I believe there is a reasonable possibility the MHS data will become identifiable | |
| @ No, I believe there is no reasonable possibility the MHS data will become identifiable | |
| 10.13 Have you completed and uploaded an appropriate HIPAA document (i.e. HIPAA Auth be obtained or Waiver/alteration of HIPAA Authorization is being requested)? ——————————————————————————————————— | orization will |
| @ Yes | |
| U No | |
| 0 N/A | |
| 10.14 Managing Data (Data Management and/or Sharing Plan) and/or Human Biological Sp<br>this Study: | ecimens for |
| Include in this section the plan for acquiring data (both electronic and hard copy), access during the study, data/specimen storage and length of time stored, shipment/transmission, and the plan for storage and final disposition at the conclusion of the study. Describe any data agreements in place for accessing data within and/or outside of your institution (e.g., Data Sharing Agreement, Data Use Agreement, Business Agreements, etc.) | |
| The consent form, baseline questionnaire, CBT outcomes, and pre-ACFT / post-ACFT self-efficacy forms will all be hard copy acquired. The post-ACFT injury case report form will be electronically acquired through Qualtrics, a secure electronic survey application. All of the case report forms (hard copy and electronic) will require the participants name on them. No subject ID will be included on these forms to remain in compliance with human research protections guidelines. Once the hard copy case report forms are collected, the study data will be transcribed into an electronic spreadsheet where the participant will only be identified by their assigned subject ID. Theonly document (electronic or hard copy) linking the subject ID and the participant name will be the electronic master subject list. The hard copy case report forms with participant names on them will all be stored together in a folder with the participant's consent form. Participant folders will be stored together in a locked filing cabinet, behind locked doors, in a CAC card protected building. All electronic files will be stored on DoD-server, CAC card protected computers. Only the PI and Al's will have access to the physical and electronic participant files. | |
| Performance information received from the Department of Military Instruction (DMI) is not | |

considered private health information, but will include personnel identifiers. The information, to include copies of ACFT scorecards, will be collected from the DMI following the ACFT and stored

with the rest of the participants hard copy CRFs containing personnel identifiers. In addition, the researchers will collect outcomes data from the DMI (CBT and task-specific event performance outcomes data) via secure access to department databases and/or via encrypted emails or an encrypted drop box.

When we are ready for data analysis, we will subsequently collect injury information, number of days on profile for each subject for up to 9 weeks following cadet basic training. Subject number of days on profile will be combined with the previously de-identified study data on a spreadsheet for analysis. The spreadsheet data will be password and firewall-protected. There are no planned linkages with external databases, nor is transmission of the data for collaborative use anticipated. The PI will keep a master spreadsheet that links subject names with their unique identification number on a government computer assigned to the PI. The computer is password and CAC-card protected, and the system is firewall protected. This document will not be shown to anyone except for the investigators in this study or governmental agencies only in accordance with federal law. All research data and forms (both paper and electronic) will only be accessible by authorized study staff, the local IRB, and applicable governmental agencies as part of their duties and in accordance with federal law. These duties include making sure that research participants are protected.

# 10.15 Managing Data (Data Management and/or Sharing Plan) and/or Human Biological Specimens for Future Research:

If the study involves collecting, storing, or banking human specimens, data, or documents (either by the Investigator or through an established repository) for FUTURE research, address. How the specimens/data will be used, where and how data/specimens will be stored (including shipping procedures, storage plan, etc.), whether and how consent will be obtained, procedures that will fulfill subjects' request as stated in the consent, whether subjects may withdraw their data/specimens from storage, whether and how subjects may be recontacted for future research and given the option to decline, whether there will be genetic testing on the specimens, who will have access to the data/specimens, and the linkage, the length of time that data/specimens will be stored and conditions under which data/specimens will be destroyed.

All records containing HIPAA PHI will be maintained for a period of 6 years at which time they will be destroyed by securely shredding. The master list connecting unique study ID to participant identifiers will be destroyed upon study closure. De-identified research data will be maintained indefinitely.

Any data submitted to an approved agency for review will be linked only to the subject identification number and not the personal identity of the participant (ie, protected health information such as name, SSN, address, phone number, etc). If the data are used in scholarly presentations or journal articles, the investigators will protect the anonymity of individual patients and will report only aggregate data (e.g. group means) where appropriate. Participants will not be specifically identified in any publication or presentation of research results. No data sharing/use agreements are necessary or will be utilized.

11.0

# Statistical/Data Analysis Plan

#### 11.1 Statistical Considerations:

List the statistical methods to be used to address the primary and secondary objectives, specific aims, and/or research hypotheses. Explain how missing data and outliers will be handled in the analysis. The analysis plan should be consistent with the study objectives. Include any subgroup analyses (e.g., gender or age group). Specify statistical methods and variables for each analysis. Describe how confounding variables will be controlled in the data analysis

To determine the effect of low back pain education (cautionary vs resiliency) on deadlift performance (weight lifted), we will use ANOVA and planned comparison analysis if between-group differences are found between groups.

To determine the effect of low back pain education on deadlift self-efficacy, we will analyze change scores with a one-way ANOVA and planned comparisons if significant.

| To determine the effect of low back pain education on perceived spine vulnerability, we will analyze change scores with a one-way ANOVA and planned comparisons if significant. | |
|---|---|
| Our study design accounts for some confounding factors by utilizing randomization. Potentially confounding variables should be balanced between groups. We will test groups at baseline to ensure they are similar among important characteristics. Furthermore, characteristics that are different among groups at baseline or that appear to be influential on load lifted will be included in the ANOVA model as a covariate to control for and test for potential confounding. | |
| 11.2 Sample Size: | |
| 1200 participants | |
| 11.3 Total number of subjects requested (including records and specimens): | |
| 1200 | |
| 11.4 If youare recruiting by study arm, please identify the arms of the study and how many sulbe enrolled in each arm N/A ———— | ojects will |
| 11.5 Please provide a justification for your sample size | |
| We have powered this study to determine a between-group difference of 5kg. This is equivalent to an effect size of d=.10 given a standard deviation of 23kg (available from previously collected data in this lab). We used G*Power 3.0 with power at .80 to calculate a total sample size of 969 subjects (323 per group). We will therefore attempt to recruit 1200 participants, allowing for 20% injury or attrition which might prevent subjects from completing the MDL event during CBT ACFT. | |
| 11.6 Data Analysis Plan: Complete description: Background, Objectives, Design, Step by Step he project is going to be done, Data analysis plan: | ow the |
| Determine if general self-efficacy is a predictor of injury during CBT by performing a Kaplan-Meier Survival Curve, a single assessment (Cadet General Self-Efficacy Assessment), analysis of the Defense Medical Surveillance System (DMSS) and a follow-up self-reported injury assessment. Independent Variable: Cadet General Self-Efficacy score Dependent Variables: Injury report according to DMSS or self-reported | |
| <ol> <li>Determine if task-specific self-efficacy is a predictor of injury during specific CBT events by performing a Kaplan-Meier Survival Curve, a single (or multiple) assessments of cadet task-specific self-efficacy, analysis of the Defense Medical Surveillance System (DMSS) and a follow-up self-reported injury assessment.</li> <li>Independent Variable: Cadet Task-Specific Self-Efficacy score</li> <li>Dependent Variables: Injury report according to DMSS or self-reported</li> </ol> | |
| 3. Determine if general self-efficacy is a predictor of performance during CBT by performing a multivariate regression between a single assessment (Cadet General Self-Efficacy Assessment) and multiple measures of performance during CBT including 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) raw or calculated score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events. 1. Independent Variable: Cadet General Self-Efficacy score 2. Dependent Variables: performance outcome by event- 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events. | |
| 4. Determine if task-specific self-efficacy is a predictor of performance during CBT by performing a multivariate regression between a single (or multiple) assessments of cadet task-specific self-efficacy, and multiple | |

measures of performance during CBT including 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) raw or calculated score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events.

- 1. Independent Variable: task-specific self-efficacy scores by event
- 2. Dependent Variables: performance outcome by event- 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events.
- 5. After completing CBT, determine which sources of self-efficacy (1) enacting mastery experiences, 2) vicarious experiences, 3) verbal persuasion, 4) physiological state, 5) affective state, 6) mental imagery) were the most influential on cadets' self-efficacy throughout CBT specific tasks including 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) raw or calculated score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events by conducting a Chi-square test.
  - 1. Independent Variable: task-specific events 1) successful completion (pass/fail), 2) Army Combat Fitness Test (ACFT) score, 3) Warrior Competition performance, 4) marksmanship score, 5) written exams, 6) swimming assessment and 7) any other individually graded events.
  - 2. Dependent Variables: reported level of influence of each (6) source of self-efficacy.
- 6. Determine the effect of low back pain education (cautionary vs resiliency) on deadlift performance (weight lifted).

We will analyze this with MDL weight lifted as the dependent variable (one-way ANOVA), with a planned comparison analysis if significant differences are found between groups.

7. Determine the degree of confidence cadets have in their ability to succeed at the MDL both before and after the education and MDL

We will analyze if there is a main effect of time in the pre-to-post self-efficacy scores with a paired I-test. We will use multiple regressions to analyze the impact of self-efficacy scores on MDL performance.

- 8. Determine the effect of low back pain education (cautionary vs resiliency) on deadlift self-efficacy. We will analyze change scores withone-way ANOVA with planned comparisons between groups if ANOVA is significant.
- 9. Determine the effect of low back pain education (cautionary vs resiliency) on perceived spine vulnerability on a deadlift.

We will analyze change scores withone-way ANOVA with planned comparisons between groups if ANOVA is significant.



# Participant Information

| 12.1 Subject Population: |
|---|
| All incoming US Military Academy cadets, class of '26, attending cadet basic training in the summer of 2022 |
| 12.2 AgeRange: |
| Check all the boxes that apply. if the age range of potential subjects (specimens, records) does not match the range(s) selected, please specify in the text box. |
| 0-17 |
| 18-24 |
| 25-34 |
| C 35-44 |
| <b>l</b> 45-54 |
| <b>1</b> 55-64 |
| C65-74 |
| <b>0</b> 75+ |
| 12.3 Gender: |

| Male |
|---|
| Female |
| Cother |
| Cottlet |
| 12.4 Special categories, check all that apply |
| C Minors /Children |
| <b>I</b> Students |
| Employees - Civilian |
| C Employees - Contractor |
| D Resident/trainee |
| Cadets / Midshipmen |
| D Active Duty Military Personnel C Wounded Warriors |
| Economically Disadvantaged Persons |
| Educationally Disadvantaged Persons |
| C Physically Challenged (Physical challenges include visual and/or auditory impairment) |
| C Persons with Impaired Decisional Capacity |
| C Prisoners |
| D Pregnant Women, Fetuses, and Neonates C Non-English Speakers |
| International Research involving Foreign Nationals - Headquarters Review is necessary |
| You must also consider the requirements of DoDI 3216.02, Enclosure 3, paragraphs 7.e. and 12. |
| 12.5 Inclusion Criteria: |
| Criteria |
| Inclusion criteria are cadets age 17-26 (cadets under the age of 18 are legally emancipated |
| 1 therefore able to consent), those paiticipating in the ACFT, and speak and understand<br>English |
| 2.1g.lo.1 |
| 12.6 Exclusion Criteria: |
| · |
| Celtoria |
| No Criteria has been added to this Protocol |
| 13.0 |
| Recruitment and Consent |
| 13.1 Please describe the recruitment process, including how subjects will be ide ntified and selected for the study. |
| -<br> |
| All 1,200 new Cadets will be recruited all together in an auditorium with a mass verbal |
| explanation and handouts available for written explanation. Researchers will be dressed in |
| professional civilian attire to prevent perceived authoritative influence due to higher military |
| rank. Cadets who do not wish to participate can decline participation. Participation is volun tary with no incentives offered for participating and those who opt out will receive no adverse actions. |

| 13.2 | Compensation for Participation: | |
|---|---|---|
| | cipation is voluntary with no incentives offered for participating and those who opt out will ve no adverse actions. | |
| 13.3 | Please describe the pre-screening process. If no pre-screening, enter Not Applicable in | the text editor |
| Not a | Not applicable | |
| 13.4 Consent Process: Revised Common Rule, Section 219.116: General requirements for informed consent, whether written or oral, are set forth in this paragraph and apply to consent obtained in accordance with the requirements set forth in paragraphs (b) through (d) of this section. Broad consent may be obtained in lieu of informed consent obtained in accordance with paragraphs (b) and (c) of this section only with respect to the storage, maintenance, and secondary research uses of identifiable private information and identifiable biospecimens. | | |
| Are y | ou requesting a waiver or alteration of informed consent? | |
| <b>0</b> Y | es ® No | |
| Pleas | se explain the consent process: | |
| Rese | archers will obtain written consent from participants all at once. | |
| 0 N | involves greater than minimal risk and recruitment of Service members occurs in a gro applicable, you may nominate an individual to serve as the ombudsman. /A opose ombudsman | |
| Prop | osed ombudsman name, if the desired ombudsman is not in the system | |
| Kelly | Channell | |
| Pleas | se explain the ombudsman's role and responsibilities on this project | |
| impa<br>He/s<br>conc<br>proce | cordance with the KACH Policy for use of an Ombudsman, the Ombudsman will act as an rtial and objective advocate for human subjects participating in research (DODI 3216.02). The will ensure that cadets are not coerced in any way and that all of their question and/or erns are answers. The Ombudsman will be present during the study recruitment and consent less to ensure voluntary involvement and that the research is presented in clear, adequate accurate means. | |
| 13.6 | Withdrawal from Study Participation: | |
| | ain the process for withdrawal and specify whether or not the subjects will be given the rtunity to withdraw their data their data/specimens in the event they wish to withdraw from study | |
| cons | articipants will receive the researchers email address during the study description and ent briefing. To be removed, they just need to email the primary investigator to be removed the study. | |

14.0

Risks and Benefits

14.1 Risks of Harm:

Identify all research-related risks of harm to which the subject **will** be exposed for each research procedure or intervention as a result of participation in this study. Consider the risks of breach of confidentiality, psychological, legal, social, and economic risks as well as physical risks. Do not describe risks from standard care procedures; only describe risks from procedures done for research purposes

The most likely risk of this study is a potential loss of privacy. We will protect subjects' privacy by labeling information only with a unique study ID number, and by keeping the link to these ID numbers in a password-protected database on a secure server which is only accessible by the principal investigator and designated research staff using CAC authentication.

There is an inherent risk of injury during cadet basic training and during the ACFT, however this study does not increase or decrease that risk. Cadets who choose to participate in this study will have identical risk as cadets who choose not to participate.

#### 14.2

### Measures to Minimize Risks of Harm (Precautions, safeguards):

For each research procedure or intervention, describe all measures to minimize and/or eliminate risk of harms to subjects and study personnel

TI1e cautionally education provided to one of the groups is similal to standat docaching advice offered to servicemembers before maximum deadlift testing or conducting an ACFT. However, in order to prevent perpetuating any participants' fear of spine vulnerability during deadlifts, we will consolidate best-evidence SIIIIIIII statements on how to maintain a healthy back as a cadet and beyond. All pa1ticipants will be given this inf01mation and provided an opportunity to speak with a licensed physical therapist about any concerns they might have about their back or lifting for the deadlift at a later date.

#### 14.3

## Confidentiality Protections (for research records, data and/or specimens):

Describe in detail the plan to maintain confidentiality of the research data, specimens, and records throughout the study and at its conclusion (e.g., destruction, long term storage, or banking). Explain the plan for securing the data (e.g., useof passwords, encryption, secure servers, firewalls, and other appropriate methods). If data will be shared electronically with other team members/collaborators outside the institution, describe the method of transmission and safeguards to maintain confidentiality. Explain whether this study may collect information that State or Federal law requires to be reported to other officials or ethically requires action, e. g., child or spouse abuse

All physical case report forms of the participants will be stored together in a locked filing cabinet which is secured behind a locked door in the Physical Therapy clinic that is located in a CAC protected building. The case report forms will be stored with the consent form of participants due to them containing personally identifiable information (first and last name).

Following the completion of data collection the study data collected on physical case report forms will be transcribed into password protected electronic spreadsheets, that will be stored on CAC protected, firewall secured, DoD server computers only accessible to the PI and AI's. The data spreadsheets will identify participants by subject ID and not by name. The master subject list is the only file that will connect subject ID and participant name.

There are no planned linkages with external databases, nor is transmission of the data for collaborative use anticipated. The PI will keep a master spreadsheet that links subject names with their unique identification number on a government computer assigned to the PI. The computer is password and CAC-card protected, and the system is firewall protected. This electronic spreadsheets will not be shown to anyone except for the investigators in this study or governmental agencies only in accordance with federal law. All research data and forms (both paper and electronic) will only be accessible by authorized study staff, the local IRB, and

applicable governmental agencies as part of their duties and in accordance with federal law. These duties include making sure that research participants are protected.

#### 14.4

#### **Potential Benefits:**

Describe any real and potential benefits of the research to the subject and any potential benefits to a specific community or society

If the individuals in the research are considered experimental subjects (per 10 USC 980), and they cannot provide their own consent, the protocol must describe the intent to directly benefit all subjects

The outcomes of this study could benefit the military community if self-efficacy proves to be an adaptable characteristic that is correlated with injury during cadet basic training. Planning training to include self-efficacy development could therefore help prevent future injury in cadets and U.S. Army Soldiers.

There is currently an emphasis in Army Doctrine {FM 7-22} on form/technique for events on the ACFT, especially the maximum deadlift (MDL) and the prevention of lower back injuries. The rationale behind this is due to the perception that breakdowns in form during the deadlift lead to injuries, however, the research does not support this. Specifically, the research is unclear regarding the position of the spine while deadlifting-neutral vs flexed. Our results could impact future DoD publications regarding technique on the MDL and deemphasize the role of a rounded spine as a safety concern.

#### 14.S

#### **Privacy for Subjects:**

Describe the measures to protect subject's privacy during recruitment, the consent process, and all research activities, etc.

Like many biomedical research protocols considered by IRBs, the protection of confidentiality is a significant concern. In order to protect confidentiality, all participants will be assigned a unique ID at the time of record review. All research related data will only be labeled and stored with each participant's unique ID. Furthermore, for the current study, only the immediate research team will have access to the data associated with this project. The linkage between the unique ID number and master participant list will be maintained electronically on the physical therapy server which is limited to authorized KACH users in the physical therapy department and requires CAC authentication.

#### 14.6

# Incidental or Unexpected Findings:

Describe the plan to address incidental findings and unexpected findings about individuals from screening to the end of the subject's participation in the research. In cases where the subject could possibly benefit medically or otherwise from the information, state whether or not the results of screening, research participation, research tests, etc., will be shared with subjects or their primary care provider. State whether the researcher is obligated or mandated to report results to appropriate military or civilian authorities and explain the potential impact on the subject

All participants will be assured that any injury information that they share with us is private and under the same protections as any other medical information. The information will not be shared with USMA administrators, faculty or cadre and will no way change the admission status or training status. We do not anticipate any unexpected findings that could be detrimental to subject. Any medical concerns will be brought up privately between the primary investigator and the cadet directly if needed.

**15.0** 

# Study Monitoring

| 15.1 Your study requires either Data and Safety Monitoring Plan (DSMP) or a Data and Safety Monitoring Board (DSMB). |
|---|
| O DSMP |
| O DOMP |
| 0 DSMB |
| O Both |
| @ Not Applicable |

16.0

## Reportable Events

16.1 Reportable Events: Consult with the research office at your institution to ensure requirements are met. Describe plans for reporting unexpected adverse events and unanticipated problems. Address how unexpected adverse events will be identified, who will report, how often adverse events and unanticipated problems will be reviewed to determine if any changes to the protocol or consent form are needed and the scale that will be used to grade the severity of the adverse event.

Consult with the research office at your institution to ensure requirements are met

- Describe plans for reporting expected adverse events. Identify what the expected adverse events will be for this study, describe the likelihood (frequency, severity, reversibility, short-term management and any long-term implications of each expected event)
- Describe plans for reporting unexpected adverse events and unanticipated problems. Address how unexpected adverse events will be identified, who will report, how often adverse events and unanticipated problems will be reviewed to determine if any changes to the research protocol or consent form are needed and the scale that will be used to grade the severity of the adverse event.

<u>Adverse events</u>: Events which are not serious are reported on the Annual Progress Report (APR) or Continuing Review Report (CRR) of the protocol.

<u>Serious Adverse Events</u>: The PI, within one working day, will report all serious adverse events occurring in participants enrolled at KACH. the investigator must contact the HPD within one business day of discovery. HPD will inform the NMCP HPD, who will notify the IRB Chair via email and phone call. The HPD will report the event to the IO as soon as possible after determining the event is an SAE or unanticipated problem. The HPD will notify DHA within 3 days that an event is under investigation and follow up by email. A Reportable Event Form and supporting documentation must be submitted to the HPD within *five* business days and will be forwarded to the IRB for review at the next available meeting.

<u>Unexpected (but not serious) adverse</u> events occurring in participants enrolled at KACH which, in the opinion of the PI, are possibly related to participation in the protocol will be reported by the PI within three working days to the IRB using the same procedure.

<u>All UPIRTSOs. UADEs, and SAEs</u> that are unexpected and determined to be at least possibly related or definitely related to research participation will be promptly reported by telephone or via email to the IRB. A complete report will follow the initial notification within three (3) business days.

Minor Deviations must be reported to the IRB at the time of continuing review or project closure.

Major Deviations should be promptly reported to the HPA and IRB and in NLT three days.

| 17.1 Does the study involve the use of any unique non-medical devices/equipment? | |
|---|---|
| O Yes @ No | |
| 18.0 FDA-Regulated Products | |
| 18.1 Will any drugs, dietary supplements, biologics, or devices be utilized in this study? | ? |
| C Drugs Dietary Supplements Biologics Devices I;i N/A | |
| 18.S Sponsor (organization/institution/company): | |
| P° N/A If applicable, provide sponsor contact information: | _ |
| Research Registration Requirements 19.1 ClinicalTrials.gov Registration: | |
| <ul> <li>Registration is not required</li> <li>Registration pending</li> <li>Registration complete</li> </ul> | |
| 19.2 Defense Technical Information Center Registration (Optional): | _ |
| <ul> <li>@ Registration is not required</li> <li>0 Registration pending</li> <li>0 Registration complete</li> </ul> | |
| 20.0 References and Glossary | |
| 20.1 References: | |
| Alemany, J. A., Pierce, J. R., Bornstein, D. B., Grier, T. L., Jones, B. H., & Glover, S. H. (2021). Comprehensive Physical Activity Assessment During U.S. Army Basic Combat Training. <i>Journal of Strength and Conditioning Research, Publish Ahead of Print.</i> https://doi.org/10.1519/JSC.0000000000004114 | |
| Almeida, P. L., Olmedilla, A., Rubio, V. J., & Palou, P. (n.d.). Psychology in the realm of sport injury: What it is all about. <i>Revista de Psicologfa Del Deporte., 23,</i> 6. | |

Army Public Health Center. (2021). *Health of the Force 2020*. Army Public Health Center. **https://phc.amedd.army.mii/ Periodical0/o20Library/ 2020-hof-report.pdf** 

Bandura, A. (2006). Guide for Construction Self-Efficacy Scales. In *Self-Efficacy Beliefs of Adolescents* (Vol. 5, pp. 307-337). Information Age Publishing.

Bandura, A. (1977). Self-efficacy: Toward a unifying theory of behavioral change. *Psychological Review*, 84(2), 191-215. https://doi.org/10.1037/0033-295X.84.2.191

Bandura, A. (1982). Self-efficacy mechanism in human agency. *American Psychologist*, 37(2), 122-147. https://doi.org/10.1037 /0003-066X.37.2.122

Beattie, S., Fakehy, M., & Woodman, T. (2014). Examining the moderating effects of time on task and task complexity on the within person self-efficacy and performance relationship. *Psychology of Sport and Exercise*, *15*(6), 605-610. https://doi.org//10.1016/j.psychsport.2014.06.007

Black, 0., Keegel, T., Sim, M. R., Collie, A., & Smith, P. (2018). The Effect of Self-Efficacy on Return-to-Work Outcomes for Workers with Psychological or Upper-Body Musculoskeletal Injuries: A Review of the Literature. *Journal of Occupational Rehabilitation*, 28(1), 16-27. https://doi.org/10.1007/s10926-017-9697-y

Brinkman, C., Baez, S. E., Genoese, F., & Hoch, J. M. (2020). Useof Goal Setting to Enhance Self-Efficacy After Sports-Related Injury: A Critically Appraised Topic. *Journal of Sport Rehabilitation*, 29(4), 498-502. https://doi.org/10.1123/jsr.2019-0032

Brouwer, S., Amick, B. C., Lee, H., Franche, R.-L., & Hogg-Johnson, S. (2015). The Predictive Validity of the Return-to-Work Self-Efficacy Scale for Return-to-Work Outcomes in Claimants with Musculoskeletal Disorders. *Journal of Occupational Rehabilitation*, 25(4), 725-732. https://doi.org/10.1007/s10926-015-9580-7

Bullock, S. H., Jones, B. H., Gilchrist, J., & Marshall, S. W. (2010). Prevention of Physical Training-Related Injuries. *American Journal of Preventive Medicine, 38(1),* 5156-5181. **https://doi.org/10.1016/j.amepre.2009.10.023** 

Center for Disease Control and Prevention/Division of Adolescent. (2020). *Trends in the Prevalence of Obesity and Dietary Behaviors, National Youth Behavior Survey 1991-2019* (p. 2). Division of Adolescent and School Health, National Center for HIV/AIDS, Viral Hepatitis, STD, and TB Prevention. <a href="https://www.cdc.gov/healthyyouth/">https://www.cdc.gov/healthyyouth/</a> data/yrbs/pdf/trends / 2019\_obesity\_trend\_yrbs.pdf

Center for Disease Control and Prevention/Division of Adolescent and School Health. (2020). *Tren ds in the Prevalence of Physical Activity and Sedentary Behaviors, National Youth Risk Behavior Survey: 1991-2019* (p. 2). Division of Adolescent and School Health, National Center for HIV /AIDS, Viral Hepatitis, STD, and TB Prevention. https://www.cdc.gov/healthyyouth/data/yrbs/pdf/trends/2019\_physical\_trend\_yrbs.pdf

Coppack, R. J., Kristensen, J., & Karageorghis, C. I. (2012). Use of a goal setting intervention to increase adherence to low back pain rehabilitation: A randomized controlled trial. *Clinical Rehabilitation*, 26(11), 1032-1042. https://doi.org/10.1177 /0269215512436613

Department of the Army. (2020). *TheU.S. Army Ho/isitic Health and Fitness Operating Concept* (p. 21). https://www.army.mil/e2/downloads/iv7 /acft/h2f\_operating\_concept.pdf

Duckworth, A. L., & Quinn, P. D. (2009). Development and Validation of the Short Grit Scale (Grit-5). *Journal of Personality Assessment*, 91(2), 166-174. https://doi.org/10.1080/00223890802634290

Dumont, G. D., Glenn, R. L., Battle, N. C., & Thier, Z. T. (2021). Correlation of the Single-Assessment Numeric Evaluation (SANE) Score With Hip-Specific Patient-Reported Outcome Measures. *Arthroscopy, Sports Medicine, and Rehabilitation*, 3(2), e435-e440. **https://doi.org/10.1016/j.asmr.2020.10.008** 

East, W.B. (2013). A Historical Review and Analysis of Army Physical Readiness Training and Assessment: Defense Technical Information Center. https://doi.org/10.21236/ ADA622014

- Feltz, D. L., Chow, G. M., & Hepler, T. J. (2008). Path Analysis of Self-Efficacy and Diving Performance Revisited. *Journal of Sport and Exercise Psychology*, *30(3)*, 401-411. **https://doi.org/ 10.1123/jsep.30.3.401**
- Gilchrist, J., Jones, B. H., Sleet, D. A., Kimsey, C. D., & CDC. (2000). Exercise-related injuries among women: Strategies for prevention from civilian and military studies. *MMWR*. *Recommendations and Reports: Morbidity and Mortality Weekly Report. Recommendations and Reports*, 49(RR-2), 15-33.
- Gilson, T. A., "Cisco Reyes, G. F., & Curnock, L. E. (2012). An Examination of Athletes' Self-Efficacy and Strength Training Effort During an Entire Off-Season. *Journal of Strength and Conditioning Research*, 26(2), 443-451.

https://doi.org/10.1519/JSC.0b013e3182254080

- Gruber, K. A., Kilcullen, R. N., & Iso-Ahola, S. E. (2009). Effects of Psychosocial Resources on Elite Soldiers' Completion of a Demanding Military Selection Program. *Military Psychology, 21(4),* 427-444. https://doi.org/10.1080/08995600903206354
- Haischer, M. H., Cooke, D. M., Carzoli, J.P., Johnson, T. K., Shipherd, A. M., Zoeller, R. F., Whitehurst, M., & Zourdos, M. C. (2021). Impact of Cognitive Measures and Sleep on Acute Squat Strength Performance and Perceptual Responses Among Well-Trained Men and Women. *Jou ma/ of Strength and Conditioning Research*, 35(1), S16-S22. https://doi.org/10.1519/JSC.000000000003202
- Hearn, D. W., Kerr, Z. Y., Wikstrom, E. A., Goss, D. L., Cameron, K. L., Marshall, S. W., & Padua, D. A. (2021). Lower Extremity Musculoskeletal Injury in USMilitary Academy Cadet Basic Training: A Survival Analysis Evaluating Sex, History of Injury, and Body Mass Index. *Orthopaedic Journal of Sports Medicine*, 9(10), 232596712110398. https://doi.org/10.1177/23259671211039841
- Helton, G. L., Cameron, K. L., Zifchock, R. A., Miller, E., Goss, D. L., Song, J., & Neary, M. T. (2019). Association Between Running Shoe Characteristics and Lower Extremity Injuries in United States Military Academy Cadets. *The American Journal of Sports Medicine*, 47(12), 2853-2862. https://doi.org/10.1177/0363546519870534
- Hutchison, A.-M., Evans, R., Bodger, O., Pallister, I., Topliss, C., Williams, P., Vannet, N., Morris, V., & Beard, D. (2013). What is the best clinical test for Achilles tendinopathy? *Foot and Ankle Surgery*, 19(2), 112-117. https://doi.org/10.1016/j.fas.2012.12.006
- Johnson, U., Tranaeus, U., & Ivarsson, A. (n.d.). Current Status and Future Challenges in Psychological Research of Sport Injury Prediction and Prevention: A Methodological Perspective. *R evista de Psico/ogia Del Deporte.*, 23, 10.
- Jones, B. H., Bovee, **M.** W., Harris, J. McA., & Cowan, D. **N.** (1993). Intrinsic risk factors for exercise-related injuries among male and female army trainees. *The American Journal of Sports Medicine*, *21*(5), 705-710. https://doi.org/10.1177/036354659302100512
- Jones, B. H., & Hauschild, V. D. (2015). Physical Training, Fitness, and Injuries: Lessons Learned From Military Studies. *Journal of Strength and Conditioning Research*, 29(Supplement 11), S57-S64. https://doi.org/10.1519/JSC.00000000001115
- Maddison, R., & Prapavessis, H. (2005). A Psychological Approach to the Prediction and Prevention of Athletic Injury. *Journal of Sport and Exercise Psychology*, 27(3), 289-310. https://doi.org/10.1123/jsep.27.3.289
- Maffulli, N., Oliva, F., Loppini, M., Aicale, R., Spiezia, F., & King, J.B. (2019). The Royal London Hospital Test for the clinical diagnosis of patellar tendinopathy. *Muscle Ligaments and Tendons Journal*, 07(02), 315. https://doi.org/10.32098/mltj.02.2017.14
- Malliaras, P., Barton, C. J., Reeves, N. D., & Langberg, H. (2013). Achilles and patellar tendinopathy loading programmes: A systematic review comparing clinical outcomes and identifying potential mechanisms for effectiveness. *Sports Medicine (Auckland, N.Z.), 43(4),* 267-286. https://doi.org/10.1007 /s40279-013-0019-z

Martinez-Calderon, J., Zamora-Campos, C., Navarro-Ledesma, S., & Luque-Suarez, A. (2018). The Role of Self-Efficacy on the Prognosis of Chronic Musculoskeletal Pain: A Systematic Review. *The Journal of Pain, 19(1),* 10-34. https://doi.org/10.1016/j.jpain.2017.08.008

Molloy, J. M. (2016). Factors Influencing Running-Related Musculoskeletal Injury Risk Among U. S. Military Recruits. *Military Medicine*, *181*(6), 512-523.

#### https://doi.org/10.7205/MILMED- D-15-00143

Molloy, J. M., Pendergrass, T. L., Lee, I. E., Chervak, M. C., Hauret, K. G., & Rhon, D. I. (2020). Musculoskeletal Injuries and United States Army Readiness Part I: Overview of Injuries and their Strategic Impact. *Military Medicine*, 185(9-10), e1461-e1471. https://doi.org/10.1093/milmed/usaa027

Molloy, J. M., Pendergrass, T. L., Lee, I. E., Hauret, K. G., Chervak, M. C., & Rhon, D. I. (2020). Musculoskeletal Injuries and United States Army Readiness. Part II: Management Challenges and Risk Mitigation Initiatives. *Military Medicine*, 185(9-10), e1472-e1480. https://doi.org/10.1093/milmed/usaa028

Moran, D. S., Evans, R., Arbel, Y., Luria, O., Hadid, A., Yanovich, R., Milgrom, C., & Finestone, A. S. (2013). Physical and psychological stressors linked with stress fractures in recruit training: Stress fractures in combat recruits. *Scandinavian Journal of Medicine & Science in Spotts*, *23(4)*, 443-450. https://doi.org/10.1111/j.1600-0838.2011.01420.x

Moran, D. S., Israeli, E., Evans, R. K., Yanovich, R., Constantini, N., Shabshin, N., Merkel, D., Luria, O., Erlich, T., Laor, A., & Finestone, A. (2008). Prediction Model for Stress Fracture in Young Female Recruits during Basic Training. *Medicine & Science in Sports & Exercise*, 40(11), S636-S644. https://doi.org/10.1249/MSS.Ob013e3181893164

Moritz, S. E., Feltz, D. L., Fahrbach, K. R., & Mack, D. E. (2000). The Relation of Self-Efficacy Measures to Sport Performance: A Meta-Analytic Review. *Research Quarterly for Exercise and Sport, 71(3), 280-294.* https://doi.org/10.1080/02701367.2000.10608908

Olmedilla, A., Rubio, V. J., Fuster-Parra, P., Pujals, C., & Garcia-Mas, A. (2018). A Bayesian Approach to Sport Injuries Likelihood: Does Player's Self-Efficacy and Environmental Factors Plays the Main Role? *Frontiers in Psychology,* 9, 1174. https://doi.org/10.3389/fpsyg. 2018.01174

Picha, K. J., Lester, M., Heebner, N. R., Abt, J.P., Usher, E. L., Capilouto, G., & Uhl, T. L. (2019). The Self-Efficacy for Home Exercise Programs Scale: Development and Psychometric Properties. *J ournal of Orthopaedic & Sports Physical Therapy*, 49(9), 647-655. https://doi.org/10.2519/jospt.2019.8779

Reiman, M., Burgi, C., Strube, E., Prue, K., Ray, K., Elliott, A., & Goode, A. (2014). The Utility of Clinical Measures for the Diagnosis of Achilles Tendon Injuries: A Systematic Review With Meta-Analysis. *Journal of Athletic Training*, 49(6), 820-829. https://doi.org/10.4085/1062-6050-49.3.36

Samendinger, S., Hill, C. R., Hepler, T. J., & Feltz, D. L. (2019). Why Residuals Are Important in the Self-Efficacy-Performance Relationship Analysis: A Study Across 12 Cycling Sessions. *Journal of Physical Activity and Health*, 16(6), 455-460. https://doi.org/10.1123/jpah.2018-0386

Samson, A. (2014). Sources of Self-Efficacy During Marathon Training: A Qualitative, Longitudinal Investigation. *The Sport Psychologist*, 28(2), 164-175.

https://doi.org/10.1123 /tsp.2013-0027

Samuels, S. M., Foster, C. A., & Lindsay, D. R. (2010). Freefall, Self-Efficacy, and Leading in Dangerous Contexts. *Military Psychology*, 22(sup1), S117-S136. https://doi.org/10.1080/08995601003644379

Shipherd, A. M., Renner, K. B., Samson, A., & Duncan, C. K. (2021). An Examination of the Sources of Self-Efficacy in Runners throughout Training: A Mixed Methods Study. 24.

Sitzmann, T., & Yeo, G. (2013). A Meta-Analytic Investigation of the Within-Person Self-Efficacy Domain: Is Self-Efficacy a Product of Past Performance or a Driver of Future Performance?: PERSONNEL PSYCHOLOGY. *Personnel Psychology*, 66(3), 531-568. https://doi.org/10.1111/peps.12035

Stasinopoulos, D., & Stasinopoulos, I. (2017). Comparison of effects of eccentric training, eccentric-concentric training, and eccentric-concentric training combined with isometric

contraction in the treatment of lateral elbow tendinopathy. *Journal of Hand Therapy, 30(1),* 13-19. https://doi.org/10.1016/j.jht.2016.09.001

Swed/er 2011 Risk Factors for Medical Discharge from BCT.pdf. (n.d.).

Swedler, D. I., Knapik, J. J., Williams, K. W., Grier, T. L., & Jones, B. H. (2011). Risk Factors for Medical Discharge From United States Army Basic Combat Training. *Military Medicine*, 176(10), 1104-1110. https://doi.org/10.7205/MILMED-D-10-00451

Taylor, S. A., & Hannafin, J. A. (2012). Evaluation and management of elbow tendinopathy. *Sport s Health*, 4(5), 384-393. https://doi.org/10.1177 / 1941738112454651

Terry, A. C., Thelen, M. D., Crowell, M., & Goss, D. L. (2018). THE MUSCULOSKELETAL READINESS SCREENING TOOL- ATHLETE CONCERN FOR INJURY & PRIOR INJURY ASSOCIATED WITH FUTURE INJURY. *International Journal of Sports Physical Therapy*, 13(4), 595-604. https://doi.org/10.26603/ijspt20180595

Thigpen, C. A., Shanley, E., Momaya, A. M., Kissenberth, M. J., Tolan, S. J., Tokish, J.M., & Hawkins, R. J. (2018). Validity and Responsiveness of the Single Alpha-numeric Evaluation for Shoulder Patients. *The American Journal of Sports Medicine*, 46(14), 3480-3485. https://doi.org/10.1177/0363546518807924

Weinberg, R. S., Gould, D., Yukelson, D., & Jackson, A. (1981). The Effect of Preexisting and Manipulated Self-efficacy on a Competitive Muscular Endurance Task. *Journal of Sport Psychology*, 3(4), 345-354. https://doi.org/10.1123/jsp.3.4.345

Adams, M.A. (1986). Hasthe lumbar spine a margin of safety in forward bending? *Clinical Biomechanics*, 1(1), 3-6. https://doi.org/10.1016/0268-0033{86})90028-8

Adams, M.A. (1994). Posture and the compressive strength of the lumbar spine. *Clinical Biomechanics*, 9(1), 10.

Arjmand, N. (2005). Biomechanics of Changes in Lumbar Posture in Static Lifting: *Spine*, 30(23), 2637-2648. https://doi.org/10.1097/01.brs.0000187907.02910.4f

Beach, T. A. C. (2018). Using verbal instructions to influence lifting mechanics - Does the directive "lift with your legs, not your back" attenuate spinal flexion? *Journal of Electromyography and Kinesiology, 38,* 1-6. https://doi.org/10.1016/j.jelekin.2017.10.008

Bengtsson, V. (2018). Narrative review of injuries in powerlifting with special reference to their association to the squat, bench press and deadlift. *BMJ Open Sport & Exercise Medicine*, 4(1), e000382. https://doi.org/10.1136/bmjsem-2018-000382

Cholewicki, J. (1991). Lumbar spine loads during the lifting of extremely heavy weights. *Medicine and Science in Sport and Exercise*, 23(10).

Cook, C. J. (2012). The effects of different pre-game motivational interventions on athlete free hormonal state and subsequent performance in professional rugby union matches. *Physiology & Behavior*, *106*(*5*), 683-688. https://doi.org/10.1016/j.physbeh.2012.05.009

Corsi, N. (2019). When words hurt: Verbal suggestion prevails over conditioning in inducing the motor nocebo effect. *European Journal of Neuroscience*, 50(8), 3311-3326. https://doi.org/10.1111/ejn.14489

Darlow, B. (2014). The development and exploratory analysis of the Back Pain Attitudes Questionnaire (Back-PAQ). *BMJ Open Sport & Exercise Medicine, 4,* 9. https://doi.org/doi: 10.1136/bmjopen-2014-005251

Dolan, P. (1994). Bending and compressive stresses acting on the lumbar spine during lifting activities. *J of Biomechanics*, 27(10), 1237-1248.

Emadi Andani, M. (2015). Modulation of Inhibitory Corticospinal Circuits Induced by a Nocebo Procedure in Motor Performance. *PLOS ONE, 10(4),* e0125223. https://doi.org/10.1371/journal.pone.0125223

Faber, G. S. (2009). Low-back loading in lifting two loads beside the body compared to lifting one load in front of the body. *Journal of Biomechanics*, 42(1), 35-41. https://doi.org/10.1016/j.jbiomech.2008.10.013

Gallagher, S. (2012). Tolerance of the lumbar spine to shear: A review and recommended exposure limits. *Clinical Biomechanics*, 27(10), 973-978. https://doi.org/10.1016/j.clinbiomech. 2012.08.009

Grimm, P. D. {2019}. Combat and Noncombat Musculoskeletal Injuries in the US Military. *Sports Medicine and Arthroscopy Review*, 27(3), 84-91. https://doi.org/10.1097/JSA. 0000000000000246

Haischer, M. H. (2021). Impact of Cognitive Measures and Sleep on Acute Squat Strength Performance and Perceptual Responses Among Well-Trained Men and Women. *Journal of Strength and Conditioning Research*, 35(1), S16-S22. https://doi.org/10.1519/JSC. 0000000000003202

Hauret, K. G. (2015). Epidemiology of Exercise- and Sports-Related Injuries in a Population of Young, Physically Active Adults: A Survey of Military Servicemembers. *The American Journal of Sports Medicine*, *43(11)*, 2645-2653. https://doi.org/10.1177/036354651560199

Hauschild, V. (2019). *Army health experts offer tips to prevent ACFT injuries*. Army.Mil. https://www.army.miljarticle/227437/army\_health\_experts\_offer\_tips\_to\_prevent\_acft\_injuries

Hendry, D. (2019). An Exploration of Pre-Professional Dancers' Beliefs of the Low Back and Dance-Specific Low Back Movements. *Medical Problems of Performing Artists*, 34(3), 147-153.

Horcajo, J. {2019). The Effects of Overt Head Movements on Physical Performance After Positive Versus Negative Self-Talk. *Journal of Sport and Exercise Psychology, 41(1),* 36-45. https://doi.org/10.1123/jsep.2018-0208

Horvath, A. {2021). Nocebo effects on motor performance: A systematic literature review. *Scandi navian Journal of Psychology*, 62(5), 665-674. https://doi.org/10.1111/sjop.12753

Jackson, Todd. (2005). The impact of threatening information about pain on coping and pain tolerance. *British Journal of Health Psychology,* 10(3), 441-451. https://doi.org/10.1348/135910705X27587

Khoddam-Khorasani, P. (2020). Effect of changes in the lumbar posture in lifting on trunk muscle and spinal loads: A combined in vivo, musculoskeletal, and finite element model study. *Journal of Biomechanics*, 104, 109728. https://doi.org/10.1016/j.jbiomech.2020.109728

Kind, L. {2019). Https://www.armytimes.com/news/your-army/2019/01/24/a-better-safer-less-expensive-alternative-to-the-new-army-pt-test/. Army Times. https://www.armytimes.com/news/your-army/2019/0 1/ 24/a-better-safer-less-expensive-alternative-to-the-new-army-pt-test/

Machida, **M.** {2017). Examining multidimensional sport-confidence in athletes and non-athlete sport performers. *Journal of Sports Sciences*, 35(5), 410-418. https://doi.org/10.1080/02640414.2016.1167934

Nolan, D. {2019}. How do manual handling advisors and physiotherapists construct their back beliefs, and do safe lifting posture beliefs influence them? *Musculoskeletal Science and Practice*, 3 9, 101-106. https://doi.org/10.1016/j.msksp.2018.11.009

Pollo, A. {2012). Preventing motor training through nocebo suggestions. *European Journal of Applied Physiology, 112(11),* 3893-3903. https://doi.org/10.1007/s00421-012-2333-9

Potvin, J. R. (1991). Trunk muscle and lumbar ligament contributions to dynamic lifts with varying degrees of trunk flexion. *Spine*, *16*(9).

Reichel, T. (2019). Incidence and characteristics of acute and overuse injuries in elite powerlifters. *Cogent Medicine*, 6(1), 1588192. https://doi.org/10.1080/233120SX.2019.1588192

Shelton, T.0. {1978). The content and effect of ?psyching-up? Strategies in weight lifters. *Cogniti ve Therapy and Research*, 2(3), 275-284. https://doi.org/10.1007/BF01185789

Sjoberg, H. (2020). Content Validity Index and Reliability of a New Protocol for Evaluation of Lifting Technique in the Powerlifting Squat and Deadlift. *Journal of Strength and Conditioning Research*, 34(9), 2528-2536. https://doi.org/10.1519/JSC.0000000000002791

Spencer, **K.** (2015). The effect of increasing loading on powerlifting movement form during the squat and deadlift. *Journal of Human Sport and Exercise*, *10(3)*. https://doi.org/10.14198/jhse. 2015.103.02

Strombiick, E. (2018). Prevalence and Consequences of Injuries in Powerlifting: A Cross-sectional Study. *Orthopaedic Journal of Sports Medicine*, 6(5), 232596711877101. https://doi.org/10.1177/2325967118771016

von Arx, M. (2021). From Stoop to Squat: A Comprehensive Analysis of Lumbar Loading Among Different Lifting Styles. *Frontiers in Bioengineering and Biotechnology*, 9, 769117. https://doi.org/10.3389/fbioe.2021.769117

Wade, K. R. (2014). How Healthy Discs Herniate: A Biomechanical and Microstructural Study Investigating the Combined Effects of Compression Rate and Flexion. *Spine*, 39(13), 1018-1028. https://doi.org/10.1097/BRS.00000000000000262

Wadey, R. (2013). Effect of Dispositional Optimism before and after Injury. *Medicine & Science in Sports & Exercise*, 45(2), 387-394. https://doi.org/10.1249/MSS.0b013e31826ea8e3

Woodman, T. (2003). The relative impact of cognitive anxiety and self-confidence upon sport performance: A meta-analysis. *Journal of Sports Sciences*, 21(6), 443-457. https://doi.org/10.1080/0264041031000101809

Zech, N. (2019). Nocebo Effects on Muscular Performance - An Experimental Study About Clinical Situations. *Frontiers in Pharmacology, 10, 219.* https://doi.org/10.3389/fphar. 2019.00219

#### 20.2 Abbreviations and Acronyms:

USMA: United States Military Academy

CBT: Cadet Basic Training MSK-I: Musculoskeletal Injury

SANE: Single Assessment Numerical Evaluation CIITS: Cadet Injury and Illness Tracking System

ACFT: Army Combat Fitness Test

MDL: Maximum Deadlift

AHLTA: Armed Forces Health Longitudinal Technology Application

DMSS: Defense Medical Surveillance System